CLINICAL TRIAL: NCT05589129
Title: Effects of a Whey Protein Supplement on Performance, Recovery, and Body Composition in Adolescent Soccer Players During the Competitive Season
Brief Title: Whey Protein Supplementation in High School Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Tanya Halliday, Principal Investigator, PhD, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 00145632
Record Dates: First submitted 2022-10-17; First posted 2022-10-21 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Body Weight Changes; Athletic Performance; Recovery; Sleep
MeSH Terms: conditions — Body Weight Changes | interventions — Whey

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Whey Protein Supplement (Experimental): Whey protein will come in powder form and will consist of 20g of protein, and 25.3g of product. We will use Optimum Nutrition Double Chocolate Whey Protein Isolate.
  Interventions: Dietary Supplement: Whey Protein Supplement
- Carbohydrate Control (Placebo Comparator): Carbohydrate control will come in powder form and will consist of 20g of carbohydrate and 21.6g of product. We will use Nesquik Chocolate Powder mix.
  Interventions: Dietary Supplement: Carbohydrate Placebo Control

INTERVENTIONS:
Dietary Supplement: Whey Protein Supplement — Participants assigned to the intervention will consume the supplement mixed with 6-8oz of water every day, twice per day, after soccer practice or soccer games, and one hour before bedtime.
  Other Names: Optimum Nutrition Gold Standard 100% Whey
  Arms: Whey Protein Supplement
Dietary Supplement: Carbohydrate Placebo Control — Participants assigned to the placebo control will consume the supplement mixed with 6-8oz of water every day, twice per day, after soccer practice or soccer games, and one hour before bedtime.
  Other Names: Nesquik Chocolate Powder
  Arms: Carbohydrate Control

SUMMARY:
The overall aim of this project is to compare protein supplementation on performance, recovery, and body composition changes in adolescent soccer players between the whey protein and the control group in response to the 10-12-week intervention.

DETAILED DESCRIPTION:
Informed Consent, Parental Permission and Assent: These will be obtained over Zoom, prior to participation in any study procedures.

Randomization: Randomization will occur following baseline testing. Participants will be randomized via random number generator stratified by sex, into either the whey protein supplement group or the placebo (isocaloric) control group.

Baseline and Post-Intervention testing will occur over a single day for each participant.

Baseline:

All athletes will report to testing facilities for a single blood draw to measure inflammatory biomarkers and a body composition assessment (via BodPod) to measure fat mass and fat free mass. Participants will then be escorted to a track where they will run a 30-yard dash to assess their speed and a 1.5-mile run to assess their estimated maximal rate of oxygen consumption (VO2max). Participants will then be transferred back to the testing facility where they will undergo assessment of lower body muscle fatigue (via HumacNorm).

Questionnaires: Athletes will complete the Munich Chronotype Questionnaire and the Pittsburg Sleep Quality Index (PSQI). Participants will also complete 3-day, 24-hour dietary recalls (via ASA-24).

Sleep measures: Fitbit (Inspire 2) will be used measure sleep efficiency, duration, and staging. Fitabase will be utilized to receive Fitbit data. Participants will be instructed to wear their Fitbit for 1-week.

Intervention:

In-season soccer practices and competition will occur 6-days per week across a 10-12 week period, depending on how far teams advance in postseason play. During the 10-12-weeks, participants will consume their assigned supplement or placebo twice per day, every day, immediately after practice or competition (or midday on rest days), and ~1 hour before bedtime.

Sleep measures: Sleep measures will be evaluated as described above. Sleep measures will be collected at weeks 2, 4, 6, 8, and 10.

Questionnaires: Participants will complete 3-days of 24-hour dietary recalls (via ASA-24) at weeks 5 and 10. Pittsburg Sleep Quality Index (PSQI), a delayed-onset muscle soreness questionnaire and a GI symptom Questionnaire will be completed at weeks 2, 4, 6, 8 and 10.

Urine Samples: We will randomly assign participants to provide urine samples at weeks 4 and 7 as a sham measure of compliance to supplementation protocol.

Post-testing will be the same as pre-testing and will commence after the 10-12-week competitive season. All measures described above in baseline testing will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* 13-18 years old; male and female High school soccer players

Exclusion Criteria:

* non-adolescents; untreated or underlying metabolic or cardiovascular diseases; allergies to dairy, or any allergies ingredients in the study provided granola bar or bagels, such as soy, wheat, tree nuts, peanuts, milk, and sesame.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Changes in Fat Free Mass | Measured at baseline and post-intervention (10-12-weeks)
  Measured via BodPod
Changes in Fat Mass | Measured at baseline and post-intervention (10-12-weeks)
  Measured via BodPod

SECONDARY OUTCOMES:
Estimated Cardiorespiratory Fitness (V02max) | Measured at baseline and post-intervention (10-12-weeks)
  Measured via 1.5-mile run time
Changes in Muscular Fatigue | Measured at baseline and post-intervention (10-12-weeks)
  Measured via leg extension machine (HumacNorm) using isometric muscle contraction in the quadriceps muscle.
Sleep Efficiency | Measured at baseline, 2-, 4-, 6-, 8-weeks and post-intervention (10-12-weeks)
  Measured via Fitbit devices. Sleep efficiency is measured based on how long and individual is asleep over the time spent in bed during the night.
Sleep Duration | Measured at baseline, 2-, 4-, 6-, 8-weeks and post-intervention (10-12-weeks)
  Measured via Fitbit devices. Sleep duration is measured based on how long the individual is asleep.
Changes in Speed | Measured at baseline and post-intervention (10-12-weeks)
  30 yard sprint
Sleep Staging | Measured at baseline, 2-, 4-, 6-, 8-weeks and post-intervention (10-12-weeks)
  Measured via Fitbit devices. Sleep stages are different periods of sleep where muscle tone and heart rate vary.

OTHER OUTCOMES:
Changes in adiponectin | Measured at baseline and post-intervention (10-12-weeks)
  Measured via blood sample to assess levels of fatty acid oxidation as well as inflammation
Changes in interleukin-6 | Measured at baseline and post-intervention (10-12-weeks)
  Measured via blood sample to assess inflammation
Changes in fibroblast growth factor 21 | Measured at baseline and post-intervention (10-12-weeks)
  Measured via blood sample to assess muscle hypertrophy
Changes in follistatin | Measured at baseline and post-intervention (10-12-weeks)
  Measured via blood sample to assess muscle hypertrophy
Changes in delayed onset muscle soreness | Measured at baseline, 2-, 4-, 6-, 8-weeks and post-intervention (10-12-weeks)
  Measured via likert scale questionnaire
Changes in Sleep quality | Measured at baseline, 2-, 4-, 6-, 8-weeks and post-intervention (10-12-weeks)
  Measured via Pittsburgh Sleep Quality Index questionnaire
Changes in dietary habits | Measured at baseline, 5-weeks and post-intervention (10-12-weeks)
  Measured via a 3-day food recall
Sleep Chronotype | Measured at baseline.
  Measured by the Munich Chronotype Questionnaire to evaluate the morningness-eveningness of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Halliday, PhD, Principal Investigator — University of Utah
Locations (1):
- Grace Zimmerman, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Request for deidentified data can be made to the PI on a case-by-case basis.